CLINICAL TRIAL: NCT07404904
Title: Evaluation of the Effects of Therapeutic Touch on Pain, Delirium, Sleep, and Physiological Parameters in Intensive Care Patients
Brief Title: Therapeutic Touch on Pain, Delirium, Sleep, and Physiological Parameters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sibel Oksuz (Other)
Collaborators: Aksaray University (Other)
Responsible Party: Sponsor-Investigator, Sibel Oksuz, Principal Investigator, Aksaray University
Organization: Aksaray University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Aksaray Hospital
Record Dates: First submitted 2025-06-18; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Sleep Disturbance; Delirium
Keywords: Therapeutic Touch; Pain; Sleep Quality; Delirium Level
MeSH Terms: conditions — Parasomnias; Delirium; Pain; Sleep Initiation and Maintenance Disorders | interventions — Therapeutic Touch

STUDY DESIGN:
Intervention Model Description: Randomized control
Who Masked: Participant
Masking Description: Participants do not know which group they are in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Randomized control (Experimental): Experimental (therapeutic touch)
  Interventions: Other: therapeutic touch
- Control (No Intervention): Control (routine care)

INTERVENTIONS:
Other: therapeutic touch — therapeutic touch
  Other Names: routine maintenance
  Arms: Randomized control

SUMMARY:
The study was conducted to determine the effects of therapeutic touch applied to intensive care patients on pain, delirium, sleep and physiological parameters.

DETAILED DESCRIPTION:
This study aims to evaluate the effects of therapeutic touch on pain, delirium, sleep, and physiological parameters in surgical intensive care patients. Patients will be assessed at 24, 48, and 72 hours. The intervention and control groups will be randomized. The intervention group will receive routine care and therapeutic touch, while the control group will receive only routine care. Parameters will be assessed before and after each measurement.

ELIGIBILITY:
Inclusion Criteria:

* Patients who volunteer to participate in the study,
* Patients aged 18 and over who receive post-surgical treatment at the Surgical Intensive Care Unit of Aksaray Education and Research Hospital,
* Patients who do not have communication problems (hearing, speaking, understanding, etc.),
* Patients who have received treatment in the surgical intensive care unit for at least 72 hours,
* Patients with RASS: between -3 and +4 and Glasgow coma scale: 10 and above,
* Patients who use only non-steroidal drugs as analgesics,
* Patients whose medical diagnosis is not dementia,
* Patients who do not have a mental state disorder/psychological disease and do not use sleeping pills.

Exclusion Criteria:

* Patients who developed complications in the ICU after surgery,
* Patients who received treatment in the surgical intensive care unit for less than 72 hours.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2024-10-10 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
VAS (Visual Analog Scale) | At 24 hours, 48 hours, and 72 hours after ICU admission (pre-intervention).
  Pain intensity measured using a 0-10 Visual Analog Scale (0 = no pain, 10 = worst pain).
RASS (Richmond Agitation and Sedation Scale) | At 24 hours, 48 hours, and 72 hours after ICU admission (pre-intervention).
  Sedation/agitation level scored from +4 (combative) to -5 (unarousable).
RCSQ (Richards-Campbell Sleep Questionnaire) | At 24 hours, 48 hours, and 72 hours after ICU admission (pre-intervention).
  Sleep quality assessed with RCSQ, range 0-100.
Blood pressure | At 24 hours, 48 hours, and 72 hours after ICU admission (pre-intervention).
  Systolic and diastolic blood pressure measured using standard bedside monitoring in the intensive care unit.
Heart rate | At 24 hours, 48 hours, and 72 hours after ICU admission (pre-intervention).
  Heart rate measured using continuous bedside cardiac monitoring in the intensive care unit.
Respiratory rate | At 24 hours, 48 hours, and 72 hours after ICU admission (pre-intervention).
  Respiratory rate measured and recorded as breaths per minute using bedside monitoring.
Body temperature | At 24 hours, 48 hours, and 72 hours after ICU admission (pre-intervention).
  Body temperature measured using a standard clinical thermometer in the intensive care unit.
Oxygen saturation | At 24 hours, 48 hours, and 72 hours after ICU admission (pre-intervention).
  Peripheral oxygen saturation measured by pulse oximetry.

SECONDARY OUTCOMES:
VAS (Visual Analog Scale) | At 24 hours, 48 hours, and 72 hours after ICU admission (post-intervention).
  Pain intensity measured using a 0-10 Visual Analog Scale.
RASS (Richmond Agitation and Sedation Scale) | At 24 hours, 48 hours, and 72 hours after ICU admission (post-intervention).
  Sedation/agitation scored from +4 to -5.
RCSQ (Richards-Campbell Sleep Questionnaire) | At 24 hours, 48 hours, and 72 hours after ICU admission (post-intervention).
  Sleep quality assessed with RCSQ, range 0-100.
Blood pressure | At 24 hours, 48 hours, and 72 hours after ICU admission (post-intervention).
  Systolic and diastolic blood pressure measured using standard bedside monitoring in the intensive care unit.
Heart rate | At 24 hours, 48 hours, and 72 hours after ICU admission (post-intervention).
  Heart rate measured using continuous bedside cardiac monitoring in the intensive care unit.
Respiratory rate | At 24 hours, 48 hours, and 72 hours after ICU admission (post-intervention).
  Respiratory rate measured and recorded as breaths per minute using bedside monitoring.
Body temperature | At 24 hours, 48 hours, and 72 hours after ICU admission (post-intervention).
  Body temperature measured using a standard clinical thermometer in the intensive care unit.
Oxygen saturation | At 24 hours, 48 hours, and 72 hours after ICU admission (post-intervention).
  Peripheral oxygen saturation measured by pulse oximetry.

CONTACTS AND LOCATIONS:
Overall Officials: Sibel Öksüz, Study Director — Aksaray University
Locations (1):
- Aksaray Universitesi, Aksaray, Turkey (Türkiye)